CLINICAL TRIAL: NCT06502600
Title: A Comprehensive Analysis of Factors Influencing Adverse Postoperative Outcomes in Hospitalized Surgical Patients
Brief Title: Factors Affecting Surgical Recovery in Hospital Patients
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2024-16-211
Record Dates: First submitted 2024-07-03; First posted 2024-07-16 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Hospitalized Surgical Patients
MeSH Terms: interventions — Operative Time; Surgeons; Operating Rooms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The favourable outcomes group
  Interventions: Procedure: surgery time; Procedure: surgeon; Procedure: surgical procedure duration; Procedure: operating room; Procedure: type of surgery
- The poor outcomes group
  Interventions: Procedure: surgery time; Procedure: surgeon; Procedure: surgical procedure duration; Procedure: operating room; Procedure: type of surgery

INTERVENTIONS:
Procedure: surgery time — This study is a retrospective observational study, with surgery time being one of the exposure factors under investigation.
Procedure: surgeon — This study is a retrospective observational study, with surgeon being one of the exposure factors under investigation.
Procedure: surgical procedure duration — This study is a retrospective observational study, with surgical procedure duration being one of the exposure factors under investigation.
Procedure: operating room — This study is a retrospective observational study, with surgical procedure duration being one of the exposure factors under investigation.
Procedure: type of surgery — This study is a retrospective observational study, with type of surgery being one of the exposure factors under investigation.

SUMMARY:
The objective of this observational study is to elucidate the factors influencing adverse postoperative outcomes in hospitalized surgical patients. The primary questions addressed are:

What factors contribute to the occurrence of adverse outcomes following surgery? How can the risks be mitigated to achieve improved postoperative outcomes?

ELIGIBILITY:
Inclusion Criteria:

* The study population consisted of all patients who had undergone surgery, with no instances of severe data missingness.

Exclusion Criteria:

* Missing data were identified where the rate of missingness was greater than 20%

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients of all inpatient surgeries conducted at a major comprehensive hospital.
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Death | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University,, Wenzhou, Zhejiang, China

REFERENCES:
- [Derived] Xie M, Zhou Z, Fei F, Deng Y, Liu C, Jin W, Chen F, Wang L, Chen C, Wang Z, Weng J, Xu Z. Risk assessment models for venous thromboembolism in surgical inpatients: a multicenter retrospective cohort study. Eur J Med Res. 2025 Nov 27;30(1):1298. doi: 10.1186/s40001-025-03575-3. PMID 41310782